CLINICAL TRIAL: NCT00862108
Title: Functional Brain Markers and Predictors of Treatment Response Associated With Norepinephrine System Genes in ADHD
Brief Title: Methylphenidate Treatment Response Study of Genetic Polymorphism in Attention Deficit Hyperactivity Disorder(ADHD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Je-Wook, Kang, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A080054
Record Dates: First submitted 2009-03-05; First posted 2009-03-16 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Polymorphism, Single Nucleotide; SLC6A2 protein, human; ADRA2A protein, human
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Methylphenidate (Experimental)
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — mg/kg dose: 0.7~1.2mg/kg PO daily morning intake 8 weeks
  Other Names: Concerta OROS; Metadate CD; Penid

SUMMARY:
The purpose of this study is to determine whether norepinephrine gene polymorphism affect to treatment response in ADHD

ELIGIBILITY:
Inclusion Criteria:

* diagnosis made by DSM-IV and K-SADS-PL
* IQ > 71

Exclusion Criteria:

* genetic disorder
* history of acquired brain injury
* seizure disorder
* other neurologic disorder
* mental disorder, pervasive developmental disorder
* obsessive-Compulsive disorder
* communication disorder
* learning disorder

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression Scale-Improvement | 8 weeks

SECONDARY OUTCOMES:
ADHD rating scale | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Churl Cho, MD, PhD, Principal Investigator — Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea